CLINICAL TRIAL: NCT01709643
Title: Postprandial Intrahepactic Lipid (IHL) and Intramyocellular Lipid (IMCL) Levels Measured With Proton Magnetic Resonance Spectroscopy (1H-MRS)
Brief Title: Postprandial IHL and IMCL Measured With Proton Magnetic Resonance Spectroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Top Institute Food and Nutrition (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: METC 12-3-025
Record Dates: First submitted 2012-10-11; First posted 2012-10-18 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2012-10

CONDITIONS: Postprandial IHL and IMCL Dynamics
MeSH Terms: interventions — Proteins

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- High fat breakfast lean subjects (Other): Subjects will consume a high fat breakfast, containing of sausage rolls. Energy content of the breakfast will be set to 50 % of the recommended daily calorie intake (BMR times 1.3).
  Interventions: Dietary Supplement: High fat breakfast
- High fat breakfast,obese subjects (Other): Subjects will consume a high fat breakfast, containing of sausage rolls. Energy content of the breakfast will be set to 50 % of the recommended daily calorie intake (BMR times 1.3).
  Interventions: Dietary Supplement: High fat breakfast
- HF breakfast with protein,lean subjects (Other): For the HFP breakfast, the subjects will consume 'Protifar' (Nutricia, Cuijk, The Netherlands) in addition to the sausage rolls. The amount of added proteins will be calculated to assure that the total energy content from proteins in the breakfast equals 20 %,
  Interventions: Dietary Supplement: HF breakfast with protein
- HF breakfast with protein,obese subjects (Other): For the HFP breakfast, the subjects will consume 'Protifar' (Nutricia, Cuijk, The Netherlands) in addition to the sausage rolls. The amount of added proteins will be calculated to assure that the total energy content from proteins in the breakfast equals 20 %,
  Interventions: Dietary Supplement: HF breakfast with protein

INTERVENTIONS:
Dietary Supplement: High fat breakfast — The HF breakfast will consist of sausage rolls ("saucijzenbroodjes"), available at the local Albert Heijn (Albert Heijn B.V., Zaandam, The Netherlands).
  Arms: High fat breakfast lean subjects; High fat breakfast,obese subjects
Dietary Supplement: HF breakfast with protein — For the HFP breakfast, the subjects will consume 'Protifar' (Nutricia, Cuijk, The Netherlands) in addition to the sausage rolls.
  Arms: HF breakfast with protein,lean subjects; HF breakfast with protein,obese subjects

SUMMARY:
The major research objective is to assess the potential of Proton Magnetic Resonance Spectroscopy to follow Intrahepatic lipid and Intramyocellular lipid dynamics after a single meal. Furthermore we aim to investigate whether the addition of protein to a high fat breakfast results in a reduced postprandial accumulation of lipids when compared to a high fat breakfast alone.

DETAILED DESCRIPTION:
Fat accumulation in non-adipose tissue, such as liver and muscle, is associated with reduced insulin sensitivity and cardiovascular disease. Little is known about the dietary determinants and the time course of this ectopic fat accumulation. Therefore the general aim of this project is to develop and validate methodology to follow postprandial hepatic and muscular lipid retention. Proton Magnetic Resonance Spectroscopy (1H-MRS) is a well-established tool for noninvasive quantification of intrahepatic lipids (IHL) and intramyocellular lipids (IMCL). Previous studies have suggested a relatively rapid regulation of IHL and IMCL levels, indicated by changes in these total lipid pools after high fat diets of 3 or 4 days. Although IHL and IMCL levels seem to change rapidly, data on IHL and IMCL levels after a single meal are lacking.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years
* Healthy
* Stable dietary habits
* No use of medication
* Lean subjects: BMI 18-25 kg/m2
* Obese subjects: BMI 30-35 kg/m2

Exclusion Criteria:

* Any medical condition requiring treatment and/or medication use
* Alcohol consumption of more than 20 g per day (± 2 units)
* Smoking
* Unstable body weight (weight gain or loss > 3 kg in the past three months)
* Participation in another biomedical study within 1 month prior to the screening visit
* Contraindications for MRI scan:

  * Central nervous system aneurysm clips
  * Implanted neural stimulator
  * Implanted cardiac pacemaker of defibrillator
  * Cochlear implant
  * Iron- containing corpora aliena in the eye or brain
  * Hearing aids and artificial (heart) valves which is contraindicated for MRS
  * Claustrophobia

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2012-09; Primary Completion 2014-06 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Difference between pre- and postprandial IHL and IMCL | 3 and 5 hours after high fat breakfast
  The primary research objective is to assess the potential of 1H-MRS to follow IHL and IMCL dynamics after a single meal in lean and obese subjects.

SECONDARY OUTCOMES:
Difference between postprandial IHL and IMCL in high fat and high fat with extra protein breakfast | 3 and 5 hours after high fat breakfast
  We aim to investigate whether the addition of protein to a high fat breakfast (HFP) results in a reduced postprandial accumulation of lipids when compared to a high fat breakfast (HF) alone.

OTHER OUTCOMES:
Fat and fat free mass of subjects | One week before the first MR measurements
  Body composition of the subjects is measured with underwaterweighing method
Blood plasma insulin levels | Ten minutes prior to high fat breakfast and 0.5, 1,2,3.5,4.5,5.5 hours after the high fat breakfast
Blood plasma glucose levels | Ten minutes prior to high fat breakfast and 0.5, 1,2,3.5,4.5,5.5 hours after the high fat breakfast
Blood plasma free fatty acid level | Ten minutes prior to high fat breakfast and 0.5, 1,2,3.5,4.5,5.5 hours after the high fat breakfast
Blood plasma triglyceride level | Ten minutes prior to high fat breakfast and 0.5, 1,2,3.5,4.5,5.5 hours after the high fat breakfast

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center +, Maastricht, Netherlands

REFERENCES:
- [Derived] Lindeboom L, Nabuurs CI, Hesselink MK, Wildberger JE, Schrauwen P, Schrauwen-Hinderling VB. Proton magnetic resonance spectroscopy reveals increased hepatic lipid content after a single high-fat meal with no additional modulation by added protein. Am J Clin Nutr. 2015 Jan;101(1):65-71. doi: 10.3945/ajcn.114.094730. Epub 2014 Nov 5. PMID 25527751